CLINICAL TRIAL: NCT03548116
Title: Biological Effects of Ultrasound Insonification of the Spleen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: John Pellerito (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor-Investigator, John Pellerito, Vice Chairman of Education, Department of Radiology; Director, Peripheral Vascular Laboratory and the Body Imaging Fellowship Program, Northwell Health
Organization: Northwell Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-0859
Record Dates: First submitted 2018-05-11; First posted 2018-06-07 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Ultrasound; Insonification; Spleen
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: After a screened individual is deemed eligible for continued participation, a study investigator will enter the participant's information into a randomization portal in order to receive the group assignment.
Who Masked: Participant, Investigator
Masking Description: The study participants will be blinded to their group assignment for the entire duration of the study. The study investigators will also be blinded to participant assignments on this study, except for the investigators performing the ultrasound procedure, co-investigators randomizing the participants, and co-investigators involved in the study's monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (7):
- Group 1 (Sham Comparator): Individuals will receive sham non-imaging mode ultrasound (control group) delivered to just the spleen's hilum (area of spleen that allows passage of blood vessels, lymphatic vessels, and nerves).
  Interventions: Device: Sham Ultrasound
- Group 2 (Experimental): Individuals will receive half-powered non-imaging mode ultrasound delivered to just the spleen's hilum (area of spleen that allows passage of blood vessels, lymphatic vessels, and nerves).
  Interventions: Device: Ultrasound
- Group 3 (Experimental): Individuals will receive full-powered non-imaging mode ultrasound delivered to just the spleen's hilum (area of spleen that allows passage of blood vessels, lymphatic vessels, and nerves).
  Interventions: Device: Ultrasound
- Group 4 (Sham Comparator): Individuals will receive sham non-imaging mode ultrasound (control group) delivered to the lower, middle, and upper spleen based on the spleen's size.
  Interventions: Device: Sham Ultrasound
- Group 5 (Experimental): Individuals will receive half-powered non-imaging mode ultrasound delivered to the lower, middle, and upper spleen based on the spleen's size.
  Interventions: Device: Ultrasound
- Group 6 (Experimental): Individuals will receive full-powered non-imaging mode ultrasound delivered to the lower, middle, and upper spleen based on the spleen's size.
  Interventions: Device: Ultrasound
- Group 7 (Sham Comparator): Individuals will receive sham non-imaging mode ultrasound with a disconnected probe (control group) delivered to just the spleen's hilum (area of spleen that allows passage of blood vessels, lymphatic vessels, and nerves).
  Interventions: Device: Sham Ultrasound

INTERVENTIONS:
Device: Ultrasound — A specially designed ultrasound will be placed against the abdomen of an individual in order to administer low levels of insonification to the spleen.
  Arms: Group 2; Group 3; Group 5; Group 6
Device: Sham Ultrasound — A specially designed ultrasound will be placed against the abdomen of an individual in order to administer sham insonification to the spleen.
  Arms: Group 1; Group 4; Group 7

SUMMARY:
This is a seven-cohort, double-blinded, randomized, sham-controlled feasibility trial to determine whether organ-specific biological effects are achievable through selective ultrasound of the spleen utilizing low-energy insonification.

DETAILED DESCRIPTION:
This study will consist of three study visits. At the screening visit, individuals will be asked to undergo a physical and neurological examination, a blood draw of 4 teaspoons, and a urine pregnancy test if of childbearing potential.

The participants that clear study screening will be randomized to one of seven groups. The groups consist of: sham insonification at the hilum (connected probe or disconnected probe); half-powered insonification at the hilum; full-powered insonification at the hilum; sham insonification at the lower, middle, and upper spleen; half-powered insonification at the lower, middle, and upper spleen; and full-powered insonification at the lower, middle, and upper spleen.

At the baseline visit, individuals will be asked to undergo a physical and neurological examination and a blood draw of 7 teaspoons before receiving ultrasound as per their assigned group. These individuals will then be asked to undergo a blood draw of 5 teaspoons at 1-hour and 2-hours after the ultrasound.

Individuals will be asked to return 24 hours later for the follow-up visit, which will include a physical and neurological examination and a blood draw of 9 teaspoons.

The blood samples collected before insonification, one hour after insonification, two hours after insonification, and twenty-four hours after insonification will be assessed for changes in biomarkers (substances in the body that indicate the status of a biological process or condition). These biomarkers include cytokines (proteins involved in the immune response), norepinephrine (chemical in the body that transmits signals), glucose (sugar in the blood), and blood cells that are involved in breathing, clotting, and the immune response.

The study will be considered complete after completion of enrollment (10 participants in each group, for a study total of 70 participants), completion of study procedures by all participants, and the completion of analysis of identifiable study data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 45 years of age
* Individuals without physical disabilities or conditions/diseases that may make them incapable of undergoing the study procedures or otherwise places them at a greater risk of harm
* Individuals without significant past medical or surgical histories that would render them at a greater risk of harm
* Individuals that are considered English Proficient due to the study requirements to follow verbal commands during the ultrasound session
* Individuals that are considered active as assessed by type of activity (i.e., walking, running, etc.) and number of hours a week performing the various activities
* Individuals able to attend all study visits at approximately the same time of day (i.e., 8 - 12 pm)
* Individuals that are able to comprehend the study goals and procedures, and are able to provide informed consent for participation

Exclusion Criteria:

* Individuals participating in another research study that may affect the conduct or results of this study
* Individuals considered substantially overweight or obese via body mass index (≥ 29)
* Individuals having or exhibiting any of the following:

  * surgery in the past 90 days
  * previous surgery of the spleen or splenectomy, esophagus, lungs, stomach, duodenum, or liver
  * recent traumatic injury, including intracerebral hemorrhage and visceral injury
  * end stage renal disease and/or uremia
  * active malignancy
  * previous leukemia and/or lymphoma
  * human immunodeficiency virus infection or AIDS
  * rheumatoid arthritis or other immune-mediated diseases (e.g. inflammatory bowel disease)
  * arrhythmias, including but not limited to, atrial fibrillation, atrial flutter, clinically significant bradycardia, ventricular arrhythmias, and A-V block
  * implanted pacemaker or cardioverter/defibrillator (AICD)
  * a history of stable or unstable angina, myocardial infarction, angioplasty or coronary arterial by-pass grafting surgery
  * history of stroke or TIA
  * history of deep venous thrombosis (DVT) and/or pulmonary embolism (PE)
  * previous episodes of pancreatitis
  * spinal disorders
  * chronic pain syndromes
  * history of thrombosis or bleeding disorders
  * stage III-IV pressure ulcers
  * sickle cell anemia or other anemia syndromes
  * monocytosis
  * thrombocytopenia
  * diagnosed with fever of unknown origin (FUO)
  * previously or currently implanted vagus nerve stimulator
  * previously or currently implanted spinal cord stimulator
  * other chronically-implanted electronic medical device
  * history of seizures
  * history of cancer
* Individuals who have taken any of the following medications within one week of receiving ultrasound delivery:

  * anti-coagulant (Coumadin, Xarelto)
  * anti-platelet (aspirin, Plavix)
  * anti-inflammatory (aspirin, NSAIDs)
  * anti-hypertensive (α-methyldopa)
  * epinephrine-related drugs, norepinephrine-related drugs, and drugs that stimulate release of epinephrine and/or norepinephrine (Micronefrin, Asthmanefrin)
  * immunosuppressive agents (steroids, newer immunomodulatory drugs)
  * alpha and/or beta adrenoceptor blocking agents
  * anti-seizure medications
  * other medications, supplements, etc. that may interfere with the ultrasound delivery or study results
* Individuals with a substance abuse (alcoholism or other) problem
* Individuals that consumed alcohol within 4 days of the baseline visit
* Individuals currently using or have used tobacco or nicotine products within the past 1 month
* Individuals currently using or have used recreational drugs within the past 1 month
* Pregnant women
* Prisoners

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Anti-inflammatory Response | The primary outcome will be assessed before ultrasound and at 1-hour, 2-hours, and 24-hours after receiving ultrasound.
  The primary outcome to determine whether diagnostic-level ultrasound to the spleen has a biological effect is measured as a statistically significant change in the level of biomarkers associated with the inflammatory response following delivery of ultrasound.

SECONDARY OUTCOMES:
Transient Tissue Displacement | The secondary outcome will be assessed approximately every 15 seconds during the approximately 10-minute ultrasound.
  The secondary outcome to determine whether ultrasound delivery to the spleen leads to transient tissue displacement that is correlated to organ-specific biological effects is measured as a statistically significant correlation between the magnitude of transient displacement and the biological effects.

CONTACTS AND LOCATIONS:
Overall Officials: John Pellerito, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health's The Feinstein Institute for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there are no plans to make individual participant data available.

REFERENCES:
- [Background] Koopman FA, Chavan SS, Miljko S, Grazio S, Sokolovic S, Schuurman PR, Mehta AD, Levine YA, Faltys M, Zitnik R, Tracey KJ, Tak PP. Vagus nerve stimulation inhibits cytokine production and attenuates disease severity in rheumatoid arthritis. Proc Natl Acad Sci U S A. 2016 Jul 19;113(29):8284-9. doi: 10.1073/pnas.1605635113. Epub 2016 Jul 5. PMID 27382171
- [Background] Zeng W, Pirzgalska RM, Pereira MM, Kubasova N, Barateiro A, Seixas E, Lu YH, Kozlova A, Voss H, Martins GG, Friedman JM, Domingos AI. Sympathetic neuro-adipose connections mediate leptin-driven lipolysis. Cell. 2015 Sep 24;163(1):84-94. doi: 10.1016/j.cell.2015.08.055. PMID 26406372
- [Background] Parker JL, Cameron T. Technology for Peripheral Nerve Stimulation. Prog Neurol Surg. 2015;29:1-19. doi: 10.1159/000434651. Epub 2015 Sep 4. PMID 26394391
- [Background] Birk DM, Yin D, Slavin KV. Regulation of Peripheral Nerve Stimulation Technology. Prog Neurol Surg. 2015;29:225-37. doi: 10.1159/000434674. Epub 2015 Sep 4. PMID 26394389
- [Background] Tracey KJ. Physiology and immunology of the cholinergic antiinflammatory pathway. J Clin Invest. 2007 Feb;117(2):289-96. doi: 10.1172/JCI30555. PMID 17273548
- [Background] Martelli D, McKinley MJ, McAllen RM. The cholinergic anti-inflammatory pathway: a critical review. Auton Neurosci. 2014 May;182:65-9. doi: 10.1016/j.autneu.2013.12.007. Epub 2013 Dec 24. PMID 24411268
- [Background] Juan EJ, Gonzalez R, Albors G, Ward MP, Irazoqui P. Vagus Nerve Modulation Using Focused Pulsed Ultrasound: Potential Applications and Preliminary Observations in a Rat. Int J Imaging Syst Technol. 2014 Mar 1;24(1):67-71. doi: 10.1002/ima.22080. PMID 25165410
- [Derived] Goggins E, Inoue H, Okusa MD. Neuroimmune Control of Inflammation in Acute Kidney Injury and Multiorgan Dysfunction. J Am Soc Nephrol. 2025 Dec 1;36(12):2473-2484. doi: 10.1681/ASN.0000000813. Epub 2025 Jul 7. PMID 40622772
- See also: Stimulating Peripheral Activity to Relieve Conditions (SPARC) — https://commonfund.nih.gov/sparc
- See also: Electrical Prescriptions — https://www.darpa.mil/program/electrical-prescriptions
- See also: Ultrasonic Stimulation of Peripheral Nervous Tissue — http://iopscience.iop.org/article/10.1088/1742-6596/581/1/012003/meta